CLINICAL TRIAL: NCT00419848
Title: the Comparison Efficacy of Azithromycin With Doxycycline in the Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Skin research center, Shaheed Beheshti Medical unversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: src-hmj-1385
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Acne
Keywords: Acne; Azithromycin; Doxycycline
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline; Azithromycin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Azithromycin
- 2 (Active Comparator)
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Cap 100mg- 100mg/daily
  Other Names: Razak lab
  Arms: 2
Drug: Azithromycin — Azithromycin: Cap 250 mg- 500 mg single dose/daily - 3 times per week
  Other Names: kimidarou
  Arms: 1

SUMMARY:
a comparison of efficacy and adverse side effects occurrence of Doxycycline and Azithromycin in the management of moderate acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Between 18 to 30 year old
* Moderate facial Acne(At least 10 inflammatory lesions with maximum 3 nodules and pseudocysts

Exclusion Criteria:

* Pregnancy
* Breast Feeding
* Acne Fulminant
* Acne conglobate
* Isotretinoin therapy within past 6 months
* topical treatment in last 2 weeks
* use of systemic antibiotic in the last month
* Hyperandrogenism symptoms
* Menstrual irregularity

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-01 (Estimated); Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
change in acne lesions | 12 weeks

SECONDARY OUTCOMES:
global response rates, patient's own assessment, side effects and compliance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Parviz Toossi, M.D., Study Chair — Skin Research Center; Hamideh Moravvej, M.D., Principal Investigator — Skin Research Center; Akbar Mousazadeh halim, M.D., Principal Investigator — Skin Research Center
Locations (1):
- Shaheed Beheshti Medical University, Skin research center, Tehran, Iran